CLINICAL TRIAL: NCT00073905
Title: Capecitabine And Gemcitabine In Patients With Advanced Or Metastatic Biliary Tract Cancer, A Multicenter Phase II Trial
Brief Title: Adjuvant Palliative Capecitabine and Gemcitabine in Treating Patients With Locally Advanced or Metastatic Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SAKK 44/02; EU-20322
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Liver Cancer; Pain
Keywords: unresectable gallbladder cancer; adenocarcinoma of the gallbladder; adenocarcinoma of the extrahepatic bile duct; unresectable extrahepatic bile duct cancer; pain; recurrent gallbladder cancer; recurrent extrahepatic bile duct cancer; localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Liver Neoplasms; Pain; Carcinoma, Hepatocellular | interventions — Capecitabine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm A (Active Comparator): Capecitabine plus Gemcitabine
  Interventions: Drug: capecitabine plus gemcitabine

INTERVENTIONS:
Drug: capecitabine plus gemcitabine — capecitabine plus gemcitabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and gemcitabine, use different ways to stop tumor cells from dividing so they stop growing or die. Palliative chemotherapy may improve the quality of life in patients who have locally advanced or metastatic biliary tract cancer and may help them live more comfortably.

PURPOSE: Phase II trial to study the effectiveness of adjuvant capecitabine and gemcitabine in improving quality of life in patients who have locally advanced or metastatic biliary tract cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the ability of palliative capecitabine and gemcitabine to maintain or improve tumor-related symptoms (after treatable biliary duct obstruction has been relieved) as measured by the clinical benefit response in patients with locally advanced or metastatic biliary tract cancer.

Secondary

* Determine the clinical benefit response in patients treated with this regimen.
* Determine the time to and duration of clinical benefit response in patients treated with this regimen.
* Determine the objective response and time to progression in patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.
* Determine the quality of life of patients treated with this regimen.
* Determine the adverse events in patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study.

Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and oral capecitabine twice daily on days 1-14 (28 total doses). Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity. Patients responding to treatment may receive additional courses at the discretion of the investigator.

Quality of life is assessed at baseline, weekly during weeks 2-9 (courses 1-3), and then before each administration of gemcitabine.

Patients are followed every 3 months for 1 year and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 19-44 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed biliary tract cancer

  * Locally advanced, unresectable, or metastatic disease
* Metastatic adenocarcinoma with clinical documentation of gallbladder or bile tree involvement with no evidence of another primary adenocarcinoma allowed
* Measurable or nonmeasurable disease
* Treatable biliary duct obstruction must be relieved by either internal endoscopic drainage/stenting or palliative bypass surgery before study entry
* Symptomatic biliary tract cancer and has at least 1 of the following:

  * Karnofsky 60-80%
  * Baseline analgesic consumption at least 10 mg of morphine equivalents per day
  * Baseline pain intensity score of at least 20 mm out of a possible 100 mm
* No prior or concurrent CNS metastasis

PATIENT CHARACTERISTICS:

Age

* 18 to 80

Performance status

* See Disease Characteristics
* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10.0 g/dL

Hepatic

* Bilirubin no greater than 4 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 5 times ULN
* AST and ALT no greater than 5 times ULN

Renal

* Creatinine clearance greater than 50 mL/min

Cardiovascular

* No uncontrolled cardiovascular disease

Gastrointestinal

* Able to ingest oral medication
* No malabsorption syndrome
* No intractable nausea and/or vomiting
* No partial small bowel obstruction

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 year after study participation
* No active autoimmune disease
* No uncontrolled diabetes
* No known hypersensitivity to fluorouracil
* No known dihydropyrimidine dehydrogenase deficiency
* No definitive contraindication to corticosteroids
* No prior significant neurologic or psychiatric disorders (e.g., psychotic disorders, dementia, or seizures) that would preclude understanding or providing informed consent
* No prior severe reaction to fluoropyrimidine therapy
* No psychiatric disorder, cognitive dysfunction, or language problem that would preclude filling out the quality of life questionnaire or patient diary
* No other serious underlying medical condition that would preclude study participation
* No other malignancy within the past 5 years except nonmelanoma skin cancer or adequately treated carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy
* No prior immunotherapy

Chemotherapy

* No prior chemotherapy for advanced/metastatic disease
* No prior palliative chemotherapy

Endocrine therapy

* No concurrent megestrol

Radiotherapy

* More than 4 weeks since prior radiotherapy
* No concurrent radiotherapy

  * Treatment of a single painful lesion allowed

Surgery

* See Disease Characteristics
* Prior Whipple procedure allowed
* Prior duodenal bypass allowed
* No concurrent endoscopic or external biliary drainage as a consequence of progressive malignant bile duct obstruction

  * Drainage as a consequence of nonmalignant bile duct obstruction allowed

Other

* More than 30 days since prior treatment within a clinical study
* No other concurrent anticancer drugs
* No other concurrent investigational drugs
* No concurrent sorivudine or its chemically-related analogues (e.g., lamivudine)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2003-04; Primary Completion 2006-06 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Ability of palliative capecitabine and gemcitabine | 3 months
  Determine the ability of palliative capecitabine and gemcitabine to maintain or improve tumor-related symptoms (after treatable biliary duct obstruction has been relieved) as measured by the clinical benefit response.

SECONDARY OUTCOMES:
Clinical benefit response alone as measured after 3 courses | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Koeberle, MD, Study Chair — Cantonal Hospital of St. Gallen
Locations (1):
- Kantonsspital - St. Gallen, Sankt Gallen, Switzerland

REFERENCES:
- [Result] Bernhard J, Dietrich D, Scheithauer W, Gerber D, Bodoky G, Ruhstaller T, Glimelius B, Bajetta E, Schuller J, Saletti P, Bauer J, Figer A, Pestalozzi BC, Kohne CH, Mingrone W, Stemmer SM, Tamas K, Kornek GV, Koeberle D, Herrmann R; Central European Cooperative Oncology Group. Clinical benefit and quality of life in patients with advanced pancreatic cancer receiving gemcitabine plus capecitabine versus gemcitabine alone: a randomized multicenter phase III clinical trial--SAKK 44/00-CECOG/PAN.1.3.001. J Clin Oncol. 2008 Aug 1;26(22):3695-701. doi: 10.1200/JCO.2007.15.6240. PMID 18669454
- [Result] Koeberle D, Saletti P, Borner M, Gerber D, Dietrich D, Caspar CB, Mingrone W, Beretta K, Strasser F, Ruhstaller T, Mora O, Herrmann R; Swiss Group for Clinical Cancer Research. Patient-reported outcomes of patients with advanced biliary tract cancers receiving gemcitabine plus capecitabine: a multicenter, phase II trial of the Swiss Group for Clinical Cancer Research. J Clin Oncol. 2008 Aug 1;26(22):3702-8. doi: 10.1200/JCO.2008.16.5704. PMID 18669455